CLINICAL TRIAL: NCT05900336
Title: Non-Steroidal Anti-Inflammatory Drug (NSAID) Response and Central Sensitization of Pain in Women With Dysmenorrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Endeavor Health (Other)
Responsible Party: Principal Investigator, Laura Payne, Assistant Professor, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2023P001489
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Dysmenorrhea; Menstrual Pain; Non-steroidal Anti-inflammatory Drug
MeSH Terms: conditions — Dysmenorrhea | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Naproxen first (Experimental): Participants take the dose of sodium naproxen during the first menstrual cycle and take the placebo during the second menstrual cycle.
  Interventions: Drug: Sodium Naproxen; Drug: Placebo
- Placebo first (Experimental): Participants take the dose of placebo during the first menstrual cycle and take the sodium naproxen during the second menstrual cycle.
  Interventions: Drug: Sodium Naproxen; Drug: Placebo

INTERVENTIONS:
Drug: Sodium Naproxen — One dose of 550mg sodium naproxen taken at the onset of at least moderate pain after menstrual bleeding has started (i.e., at least 6/10 on the 0-10 numeric rating scale).
Drug: Placebo — One dose of placebo capsule taken at the onset of at least moderate pain after menstrual bleeding has started (i.e., at least 6/10 on the 0-10 numeric rating scale).

SUMMARY:
Menstrual pain is the most common gynecological complaint and the leading cause of school and work absences in reproductive-age girls and women. One of the primary treatments for menstrual pain is use of nonsteroidal anti-inflammatory drugs (NSAIDs; over-the-counter medications such as naproxen, ibuprofen, or aspirin), although up to 18% of women do not get pain relief from these medications. One reason for this may be due to central sensitization of pain, which is when alterations in the central nervous system change how pain is processed in the brain and experienced. Determining the role of central sensitization in menstrual pain is important because central sensitization is associated with the development of chronic pain. Understanding the relationship between NSAID response and central sensitization is important because it could indicate women who may go on to develop chronic pain later in life. This study would directly address this question. Identifying women at risk for chronic pain would help target new treatments to this vulnerable group to ideally prevent pain from becoming chronic. This is particularly important for women in the military because the severity of menstrual pain is associated with missed work, such that in active-duty military women, less than 4.4% with mild menstrual pain missed work, whereas 20.7% of women with moderate to severe menstrual pain missed work. Addressing the significant impact of menstrual pain for military women will help reducing suffering and potentially decrease the risk of developing future chronic pain problems in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18-50 years
2. Menstrual pain rated at least 6/10 on a 0 (no pain) to 10 (worst pain possible) NRS for all menstrual cycles in the previous 6 months
3. Regular menstrual cycles over the past year (at least 9 in the previous 12 months)
4. Self-reported menstrual cycle averaging 22-35 days
5. Access to a smartphone and email, and willing/able to receive text messages
6. Able to read and understand English
7. Ability and willingness to provide written informed consent.

Exclusion Criteria:

1. Use of oral contraceptives or any exogenous hormones in the previous 3 months prior to participation
2. Variable levels of menstrual pain in the previous 6 months
3. Self-reported symptoms consistent with a chronic pain condition (e.g., pain in any body area lasting longer than 3 months) or previous diagnosis of a chronic pain condition
4. Currently pregnant or breastfeeding
5. History of pelvic inflammatory disease or sexually transmitted disease
6. Acute illness or injury that would potentially impact pain task performance (e.g., fever, flu symptoms) or that affect sensitivity of the extremities (e.g., Reynaud's disease)
7. Allergy to naproxen or having a health condition that contradicts use of naproxen or affects naproxen metabolism (e.g., kidney disease)
8. History of high blood pressure or anemia (due to possible complications from NSAID use).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Overall NSAID response | 4 hrs after taking dose during the 2nd medicated menstrual period (i.e., 4 hrs after the first occurrence of pain >= 6 on the 0-10 scale after menstrual bleeding has started during the 2nd medicated menstrual period); # of days varies by participant
  NSAID response will be calculated by comparing change in menstrual pain ratings following NSAID to change in menstrual pain ratings following placebo. Calculated by subtracting the placebo cycle response measure from the NSAID cycle response measure. This will result in a single measure indicative of the degree of NSAID response, while controlling for placebo effects
Urinary naproxen concentration | Four hours after taking the dose (either Naproxen or placebo).
  Concentration of naproxen measured in the urine sample.
Conditioned pain modulation (CPM) | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  Conditioned pain modulation (CPM) assesses pain inhibition. CPM is calculated as the change in pain50 between when the pressure is applied by itself (test stimulus) and when it is applied while the participant's hand is submerged in cold water (conditioning stimulus).

SECONDARY OUTCOMES:
Placebo cycle response | 4 hours after dose is taken.
  Change in menstrual pain rating on a 0 (no pain) to 10 (worst pain possible) numeric rating scale before and after the dose is taken. Calculated by subtracting the pre-dose rating from the post-dose rating.
NSAID cycle response | 4 hours after dose is taken.
  Change in menstrual pain rating on a 0 (no pain) to 10 (worst pain possible) numeric rating scale before and after the dose is taken. Calculated by subtracting the pre-dose rating from the post-dose rating.
Urinary PGF2α concentration | Four hours after taking the dose (either Naproxen or placebo).
  Concentration of prostaglandin F2α (PGF2α) measured in the urine sample.
Urinary PGE concentration | Four hours after taking the dose (either Naproxen or placebo).
  Concentration of prostaglandin E (PGE) measured in the urine sample.
pain50 | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The amount of pressure in kg/cm2 at the first instance of a pain rating of at least 50/100 during an ascending series of 5-second pressures applied to the dominant thumbnail. [Pressures begin at 0.5 kg/cm2 and increase by steps of 0.5 kg/cm2. The pressure sequence is terminated when the participant reaches their individual tolerance and decides to stop, when the participant reaches the safety maximum amount of pressure, or when the participant rates the pressure >=70 on a 0 (no pain) to 100 (worst pain possible) numeric rating scale.]
pain70 | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The amount of pressure in kg/cm2 at the first instance of a pain rating of at least 70/100 during an ascending series of 5-second pressures applied to the dominant thumbnail. [Pressures begin at 0.5 kg/cm2 and increase by steps of 0.5 kg/cm2. The pressure sequence is terminated when the participant reaches their individual tolerance and decides to stop, when the participant reaches the safety maximum amount of pressure, or when the participant rates the pressure >=70 on a 0 (no pain) to 100 (worst pain possible) numeric rating scale.]
Pressure pain sensitivity (PPS) | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The pain rating [on a 0 (no pain) to 100 (worst pain possible) numeric rating scale] of a 5-second, 2.0 kg/cm2 application of pressure to the dominant thumbnail bed.
Pressure pain tolerance (PPT) | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The last rated pressure delivered in a series of increasing pressure applications to the right thumbnail bed. Each application of pressure lasts for 5 seconds. The pressure sequence is terminated when the participant reaches their individual tolerance and decides to stop, when the participant reaches the safety maximum amount of pressure, or when the participant rates the pressure >=70 on a 0 (no pain) to 100 (worst pain possible) numeric rating scale.
Trapezius pressure pain sensitivity (TPPS) | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The pain rating [on a 0 (no pain) to 100 (worst pain possible) numeric rating scale] of a 5-second, 4.0 kg/cm2 application of pressure to the dominant trapezius muscle.
Time to bladder first sensation | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The amount of time in minutes from when the participant began drinking water during the bladder pain task to when she first feels able to urinate.
Pain at bladder first sensation | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The amount of bladder pain rated on a 0 (no pain) to 100 (worst pain possible) during the bladder pain task when the participant first feels able to urinate.
Time to bladder first urge | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The amount of time in minutes from when the participant began drinking water during the bladder pain task to when she reaches a point at which she would request to use the restroom if participating in an activity.
Pain at bladder first urge | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The amount of bladder pain rated on a 0 (no pain) to 100 (worst pain possible) during the bladder pain task when the participant reaches a point at which she would request to use the restroom if participating in an activity.
Time to bladder maximum tolerance | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The amount of time in minutes from when the participant began drinking water during the bladder pain task to when she is no longer able to hold more urine.
Pain at bladder maximum tolerance | At baseline (i.e., during the in-person study visit, during days 8-14 of the menstrual cycle, prior to either of the medication cycles)
  The amount of bladder pain rated on a 0 (no pain) to 100 (worst pain possible) during the bladder pain task when the participant is no longer able to hold more urine.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Payne, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No